CLINICAL TRIAL: NCT00747565
Title: Clinical Evaluation of the Tecnis Multifocal Intraocular Lens (IOL), Model ZM900, Original Study (DIOL-101-TCNS); Clinical Evaluation of the Tecnis Multifocal Intraocular Lens, Model ZM900, Expansion Study (DIOL-104-TCNS)
Brief Title: Safety and Effectiveness of a Multifocal Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIOL-104-TCNS & DIOL-101-TCNS
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: cataract, tecnis, multifocal, intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecnis Multifocal IOL group (Experimental): Subjects implanted bilaterally with the Tecnis Multifocal IOL. Participants were enrolled in this arm in the original study and also in the expansion study. Outcomes of the first eye of each subject were analyzed for the primary study endpoints.
  Interventions: Device: Tecnis ZM900 Multifocal Intraocular Lens
- CeeOn 911A monofocal control IOL group (Active Comparator): Subjects implanted bilaterally with the CeeOn 911A monofocal IOL. Participants enrolled in this arm only in the original study; no control subjects were enrolled in the expansion study. Outcomes of the first eye of each subject were analyzed for the primary study endpoints.
  Interventions: Device: CeeOn 911A monofocal IOL

INTERVENTIONS:
Device: Tecnis ZM900 Multifocal Intraocular Lens — Investigational intraocular lens
  Arms: Tecnis Multifocal IOL group
Device: CeeOn 911A monofocal IOL — Monofocal Control IOL
  Arms: CeeOn 911A monofocal control IOL group

SUMMARY:
To evaluate the safety and effectiveness of the ZM900 Tecnis Multifocal lens. Results from two studies (an original study with 125 multifocal and 123 monofocal subjects, protocol DIOL-101-TCNS, and an expansion study with 222 additional multifocal subjects, protocol DIOL-104-TCNS) are combined to evaluate the ZM900 Tecnis Multifocal lens vs. a monofocal control. The original study was conducted in 2004-2006; the expansion study was conducted in 2007-2008. Results from both studies were analyzed together for FDA approval.

DETAILED DESCRIPTION:
The original study was protocol DIOL-101-TCNS; the expansion study was protocol DIOL-104-TCNS. The study protocols were almost identical with the exception that no control subjects were enrolled in the expansion study; only additional multifocal subjects. All eligibility criteria and testing conducted in the expansion study was the same as that in the original study. The hypotheses were that best corrected distance visual acuity of the ZM900 lens would meet or exceed the FDA grid values, complication and adverse event rates of the ZM900 would be similar to the FDA grid rates for posterior chamber IOLs, and near visual acuity of the ZM900 lens would be improved compared to that of the monofocal control lens.

ELIGIBILITY:
Inclusion Criteria:

* Visual potential of 20/30 or better in each study eye
* Preoperative BCDVA worse than Snellen 20/40 or worse than 20/30 in the presence of glare (as measured using a Snellen chart with BAT at medium)
* Naturally dilated pupil size (in dim light) > 4.0 mm (with no dilation medications) for each study eye
* Preoperative corneal astigmatism of 1.0 D or less

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision (the use of any miotic agent is specifically contraindicated)
* Acute or chronic disease or illness that would increase the operative risk or confound the study outcome(s),(e.g., diabetes mellitus, immunocompromised, connective tissue disease, etc.)
* Uncontrolled systemic or ocular disease
* History of ocular trauma or prior ocular surgery or subjects expected to require retinal laser treatment or other surgical intervention
* Presence of ocular pathology other than cataract such as:

  * Amblyopia or strabismus
  * Corneal abnormalities
  * Pupil abnormalities
  * Capsule or zonule abnormalities
  * Intraocular inflammation
  * Known pathology that may affect visual acuity and/or are predicted to cause future acuity losses to a level of 20/30 or worse (e.g. macular degeneration)
* Requiring an intraocular lens outside the study diopter range
* Contact lens usage prior to study procedure (time interval dependent upon contact lens type)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2004-11; Primary Completion 2008-01 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, M.D., Principal Investigator — Drs. Fine, Hoffman and Packer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multifocal and monofocal control subjects were enrolled in the original study in 2004-2005 from the normal cataract populations at 13 USA sites. In the expansion study, additional multifocal subjects were enrolled from the normal cataract populations at 16 USA sites (13 who also participated in the original study) in 2007.
Pre-assignment Details: Subjects chose which type of lens to receive (multifocal or monofocal) in the original study. Subjects only received the multifocal lens in the expansion study.
Groups:
- Tecnis Multifocal Subjects: Note: only outcomes of the first eye implanted of each Tecnis Multifocal subject were analyzed for primary endpoints.
- Monofocal Control Subjects: Note: Only outcomes of the first eye implanted of each monofocal control subject were analyzed for primary endpoints.
Period: Overall Study
Arm/Group | Tecnis Multifocal Subjects | Monofocal Control Subjects
Started | 347 (125 multifocal subjects in original study plus 222 multifocal subjects in the expansion study.) | 123
Completed | 333 (118 multifocal subjects in the original study plus 215 multifocal subejcts in the expansion study.) | 116
Not Completed | 14 | 7
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecnis Multifocal Subjects | Monofocal Control Subjects | Total
Number analyzed (Participants) | 347 | 123 | 470
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 144 | 27 | 171
  >=65 years | 203 | 96 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.5) | 68.7 (8.9) | 66.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 81 | 292
  Male | 136 | 42 | 178
Region of Enrollment [Number; unit: participants]
  United States | 347 | 123 | 470

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieved Best Corrected Distance Visual Acuity of 20/40 or Better in the First Eye.
Description: Number of participants that achieved a best corrected distance visual acuity of 20/40 or better in the first eye. As most subjects were implanted bilaterally,"first eye" refers to the first implanted eye of each subject.
Time Frame: One year
Population: First eye results from subjects at one year in both the original study and the expansion study combined.
Measure: Number; unit: Participants (First Eyes only)
Arm/Group | Tecnis Multifocal Subjects | Monofocal Control Subjects
Number analyzed (Participants) | 331 | 114
Participants (First Eyes only) | 329 | 114

2. Primary Outcome: Mean Binocular Distance Corrected Near Visual Acuity in Snellen
Description: Mean binocular near visual acuity with distance correction in place measured at 33 cm; Mean is reported in Snellen (e.g. 20/20, 20/40, etc.), standard deviation reported in ETDRS (Early treatment diabetic retinopathy study)eye chart log units.
Time Frame: One year
Population: Binocular subjects at one year available for testing for both studies combined.
Measure: Mean (Standard Deviation); unit: Mean Snellen Line (with ETDRS line SD)
Arm/Group | Tecnis Multifocal Subjects | Monofocal Control Subjects
Number analyzed (Participants) | 291 | 113
Mean Snellen Line (with ETDRS line SD) | 24 (1.09) | 70 (1.64)
Statistical Analysis 1: Comparison: Tecnis Multifocal Subjects vs Monofocal Control Subjects; ETDRS line scores used for statistical comparisons with mean Snellen values reported above; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Tecnis Multifocal Subjects: Note: only outcomes of the first eye implanted of each Tecnis Multifocal subject were analyzed for primary endpoints. One additional multifocal subject was enrolled but received an incorrect lens; this subject is included for adverse event reporting for a total of 348 (347 +1) multifocal subjects.
Arm/Group | Tecnis Multifocal Subjects | Monofocal Control Subjects
Serious Adverse Events (participants affected / at risk) | 14/348 | 1/123
Other Adverse Events (participants affected / at risk) | 0/348 | 0/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecnis Multifocal Subjects (N=348) | Monofocal Control Subjects (N=123)
Endophthalmitis, hypopyon and surgical intervention (Eye disorders) | 1 (5) | 0 (0)
Signifcant loss in vision due to stroke (Eye disorders) | 1 (1) | 0 (0)
Lens-related lens removal (Eye disorders) | 1 (1) | 0 (0)
Lens-related other surgical procedures (Eye disorders) | 1 (1) | 0 (0)
Non-lens-related lens exchange (Eye disorders) | 4 (4) | 0 (0)
Non-lens-related other surgical procedures (Eye disorders) | 6 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
Results from the original study (DIOL-101-TCNS) and the expansion study (DIOL-104-TCNS) were analyzed together. The original study enrolled both multifocal and monofocal control subjects; the expansion study enrolled additional multifocal subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may not publish or disclose study data without Sponsor's prior written approval.